CLINICAL TRIAL: NCT06570889
Title: VItamin D in pregnanCy for prevenTion Of eaRlY Childhood Asthma (VICTORY)
Brief Title: VItamin D in pregnanCy for prevenTion Of eaRlY Childhood Asthma
Acronym: VICTORY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Klaus Bønnelykke (Other)
Responsible Party: Sponsor-Investigator, Professor Klaus Bønnelykke, Professor PhD, Head of COPSAC, Copenhagen Studies on Asthma in Childhood
Organization: Copenhagen Studies on Asthma in Childhood (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-23055833-D
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Asthma; Respiratory Tract Infections; Gastrointestinal Infection; Croup; Eczema; Allergy; Wheezing; Fractures, Bone; Development, Child; Cognition Disorders in Children; Psychiatric Diagnosis
Keywords: Childhood; Asthma; Infections; Eczema; Allergy; Development; Psychiatry; Bone development; Cognition; Growth
MeSH Terms: conditions — Asthma; Respiratory Tract Infections; Croup; Eczema; Hypersensitivity; Respiratory Sounds; Fractures, Bone; Mental Disorders; Infections | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 (cholecalciferol) 3200 IU/day (Experimental): Oral intake of 1 capsule daily from week 22-26 of gestation until 1 week after delivery
  Interventions: Dietary Supplement: Cholecalciferol D3
- Placebo Pearls with olive oil (Placebo Comparator): Oral intake of 1 capsule daily from week 22-26 of gestation until 1 week after delivery
  Interventions: Other: Olive oil

INTERVENTIONS:
Dietary Supplement: Cholecalciferol D3 — Oral intake of 1 capsule per day from week 22-26 in pregnancy to 1 week after delivery
  Other Names: D-Pearls, PharmaNord, DK
  Arms: Vitamin D3 (cholecalciferol) 3200 IU/day
Other: Olive oil — Oral intake of 1 capsule per day from week 22-26 in pregnancy to 1 week after delivery
  Other Names: Placebo Pearls, PharmaNord, DK
  Arms: Placebo Pearls with olive oil

SUMMARY:
The overall aim of the study is to develop a nutritional preventive vitamin D supplementation strategy in pregnancy for early childhood asthma/persistent wheeze during the first three years of life as we hypothesize that supplementation in higher doses than recommended could reduce the risk of disease development.

DETAILED DESCRIPTION:
Randomization of 2000 pregnant women to vitamin D of high-dose (3200 IU/day) vitamin D vs placebo on top of the recommended 400 IU/day. Supplementation begins in gestational week 24 (22-26) until 1 week after delivery. Allocation to the trial will be determined based on the pre-interventional maternal blood levels of EPA+DHA with a dried blood screening test. Women with high levels (above 4.7% of total fatty acids) will be assigned to the vitamin D RCT. Maternal blood will be used for genetic, metabolomic and proteomic profiling. A 3-year follow-up of the children with longitudinal registration of parent reported symptoms, diagnoses, medication use, and hospitalizations will be performed. The primary outcome is persistent wheeze or asthma until age 3 years, with predefined analyses of effect modification by maternal genotypes. Secondary outcomes are lower respiratory tract infections, gastrointestinal infections, croup, troublesome lung symptoms, eczema, allergy, bone fractures, developmental milestones, mental health, cognition, and growth until age 3 years. A follow-up on both primary and secondary outcomes is planned after unblinding, from age 3 to 6 years.

ELIGIBILITY:
* Pregnant Danish women before week 26 with blood levels of EPA+DHA above 4.7% of total fatty acids
* No current vitamin D intake above the recommended 400 IU/day
* No endocrine-, heart-, kidney- or auto-immune disorders
* No disorders requiring treatment with blood thinning medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Early childhood asthma/persistent wheeze age 0-3 years | 3 years
  Defined as either a) parental report of a minimum of 2 wheeze episodes with at least 1 after the child's second birthday and redemption of at least 2 prescriptions of asthma controller medication with at least 1 being after the child's second birthday or b) a minimum of 2 ED visits or hospitalizations due to asthmatic symptoms, and at least 1 of these being after the child's second birthday or c) parental report of physician-diagnosed asthma age 0-3 years
  Outcome analysis: risk (survival analysis) of persistent wheeze or asthma at age 0-3 years.

SECONDARY OUTCOMES:
Atopic/non-atopic wheeze or asthma age 0-3 years | 3 years
  Parental reports of physician diagnosed asthma in combination with eczema and/or allergic rhinitis.
  Outcome analyses: asthma/persistent wheeze with/without eczema and/or allergic rhinitis (yes/no) by age 3 years. Each subtype is compared with children without asthma.
Troublesome lung symptoms age 0-3 years | 3 years
  Defined as cough, wheeze or dyspnea severely affecting the well-being of the child for at least 3 consecutive days based on parental reports.
  Outcome analyses: total no. of episodes with symptoms age 0-3 years.
Wheeze episodes age 0-3 years | 3 years
  Parental reports of wheezing. Outcome analyses: total no. of episodes with wheeze age 0-3 years.
Inhaled bronchodilator use from parental reports age 0-3 years | 3 years
  Outcome analyses: total no. of days with bronchodilator use age 0-3.
Inhaled bronchodilator prescriptions from medical record checks age 0-3 years | 3 years
  Outcome analyses: total no. of prescriptions age 0-3.
Asthma controller medication use from parental reports age 0-3 years | 3 years
  Outcome analyses: total no. of days with use of asthma controller medication age 0-3.
Asthma controller medication prescriptions from medical record checks age 0-3 years | 3 years
  Outcome analyses: total no. of prescriptions age 0-3.
Asthma hospitalizations or emergency department visits age 0-3 years | 3 years
  Outcome analyses: total no. of episodes age 0-3 years.
Eczema age 0-3 years | 3 years
  Parental reports of physician-diagnosed eczema and prescribed topical antiinflammatory medication on medical record checks.
  Outcome analyses: risk (survival analysis) of any eczema age 0-3 years and current eczema (yes/no) by age 3 years.
Allergic rhinitis age 0-3 years | 3 years
  Based on parental reports of physician-diagnosed allergic rhinitis.
  Outcome analyses: allergic rhinitis (yes/no) by age 3 years.
Food allergy 0-3 years | 3 years
  Parental reports of physician-diagnosed food allergy.
  Outcome analyses: any food allergy (yes/no) by age 3 years.
Lower respiratory tract infections age 0-3 years | 3 years
  Parental reports of physician-diagnosed bronchiolitis or pneumonia.
  Outcome analysis: risk (survival analysis) of first lower respiratory tract infection and total no. of lower respiratory tract infections age 0-3 years.
Gastrointestinal infections age 0-3 years | 3 years
  Parental reports.
  Outcome analyses: risk (survival analysis) of any gastroenteritis episode and total no. of gastroenteritis episodes age 0-3 years.
Croup age 0-3 years | 3 years
  Parental reports of physician diagnosed croup.
  Outcome analysis: risk (survival analysis) of any croup episode and total no. of croup episodes age 0-3 years.
Fever episodes age 0-3 years | 3 years
  Based on parental reports.
  Outcome analyses: total no. of episodes with symptoms age 0-3 years.
Absences from daycare age 0-3 years | 3 years
  Due to illnesses based on parental reports.
  Outcome analyses: total no. of absence days age 0-3 years.
Bone fractures age 0-3 years | 3 years
  Assessed by medical record checks including all radiologically verified fractures of larger long bones (i.e. clavicle, radius, ulna, tibia, fibula, femur and humerus).
  Outcome analyses: total no. of fractures age 0-3 years.
Developmental milestones age 0-3 years | 3 years
  Monitored every 6 months until age 3 years by the parents using a registration form based on The Denver Development Index and WHO milestones registration.
  Outcome analyses: combined assessment of age at achievement across milestones by principal component analysis.
Strength and difficulties at age 3 years | 3 years
  From the Strengths and Difficulties Questionnaire (SDQ), which is a brief behavioral screening questionnaire.
  Emotional symptoms: range 0-10, a low score means better outcome. Behavioral symptoms: range 0-10, a low score means better outcome. Hyperactivity/attention difficulties:range 0-10, a low score means better outcome.
  Problems with children of the same age:range 0-10, a low score means better outcome.
  Social strengths:range 0-10, a high score means better outcome. Impact on well-being and functioning: range 0-10, a low score means better outcome.
  Outcome analyses: SDQ scores at age 3 years.
BMI age 0-3 years | 3 years
  From parental reports every 6 months.
  Outcome analyses: development of BMI age 0-3 years and current BMI at age 3.
Waist circumference age 0-3 years | 3 years
  From parental reports every 6 months.
  Outcome analyses: development of waist circumference age 0-3 years and current waist circumference at age 3.
Persistent wheeze or asthma age 0-6 years | 6 years
  Defined similarly to the primary outcome
  Outcome analysis: risk (survival analysis) of persistent wheeze or asthma at age 0-6 years
Current asthma at age 6 years | 6 years
  Defined similarly to the primary outcome and with symptoms and/or asthma medication use in the last 12 months at age 6.
  Outcome analyses: Current wheeze or asthma (yes/no) by age 6 years.
Asthma or wheeze yearly prevalence 0-6 years | 6 years
  Defined as in the primary outcome and current disease defined from parental reports of wheeze and/or asthma medication use.
  Outcome analyses: Yearly prevalence of wheeze or asthma medication use (yes/no) 0-6 years.
Atopic/non-atopic asthma at age 6 years | 6 years
  Parental reports of physician diagnosed asthma in combination with eczema and/or allergic rhinitis.
  Outcome analyses: Current asthma with/without eczema and/or allergic rhinitis (yes/no) by age 6 years. Each subtype is compared with children without asthma.
Asthma controller medication 0-6 years | 6 years
  From redeemed medication prescriptions (inhaled corticosteroids and leukotriene modifiers) based on medical record checks:
  Outcome analyses: total no. of prescriptions age 0-6 years.
Inhaled bronchodilators age 0-6 years | 6 years
  From redeemed inhaled bronchodilators based on medical record checks.
  Outcome analyses: total no. of prescriptions age 0-6 years.
Asthma hospitalizations or emergency department visits age 0-6 years | 6 years
  Based on medical record checks.
  Outcome analyses: total no. of episodes age 0-6 years.
Eczema age 0-6 years | 6 years
  Based on parental reports of physician diagnosed eczema.
  Outcome analyses: risk (survival analysis) of any eczema age 0-6 years and current eczema (yes/no) by age 6 years.
Allergic rhinitis age 0-6 years | 6 years
  Based on parental reports of physician-diagnosed allergic rhinitis and on medical record checks.
  Outcome analyses: allergic rhinitis (yes/no) by age 6 years.
Food allergy age 0-6 years | 6 years
  Based on parental reports of physician-diagnosed food allergy.
  Outcome analyses: any food allergy (yes/no) by age 6 years.
Lower respiratory tract infections age 0-6 years | 6 years
  Based on parental reports of physician-diagnosed bronchiolitis or pneumonia.
  Outcome analysis: risk (survival analysis) of first lower respiratory tract infection and total no. of lower respiratory tract infections age 0-6 years.
Gastrointestinal infections age 0-6 years | 6 years
  Based on parental reports.
  Outcome analyses: risk (survival analysis) of any gastroenteritis episode and total no. of gastroenteritis episodes age 0-6 years.
Croup age 0-6 years | 6 years
  Based on parental reports of physician diagnosed croup.
  Outcome analysis: risk (survival analysis) of any croup episode and total no. of croup episodes age 0-6 years.
Bone fractures age 0-6 years | 6 years
  Assessed by medical record checks including all radiologically verified fractures of larger long bones (i.e. clavicle, radius, ulna, tibia, fibula, femur and humerus).
  Outcome analyses: total no. of fractures age 0-6 years.
Strength and difficulties at age 6 years | 6 years
  From the Strengths and Difficulties Questionnaire (SDQ), which is a brief behavioral screening questionnaire.
  Emotional symptoms: range 0-10, a low score means better outcome. Behavioral symptoms: range 0-10, a low score means better outcome. Hyperactivity/attention difficulties:range 0-10, a low score means better outcome.
  Problems with children of the same age:range 0-10, a low score means better outcome.
  Social strengths:range 0-10, a high score means better outcome. Impact on well-being and functioning: range 0-10, a low score means better outcome.
  Outcome analyses: SDQ scores at age 6 years.
ADHD symptoms at age 6 years | 6 years
  From the ADHD rating scale-IV preschool, a dimensional questionnaire for ADHD symptoms in preschool children.
  For attention symptoms: range: 0-27, a low score means better outcome. For impulsivity-hyperactivity: range: 0-27, a low score means better outcome. For behavioral problems: range: 0-24, a low score means better outcome.
  Outcome analyses: ADHD symptom scores at age 6 years.
Psychopathology screening at age 6 years | 6 years
  From the Child Behavior Check List; a questionnaire for general screening of preschool psychopathology.
  Total problem score: range 0-236, a low score means better outcome Internalizing problems score: range 0-64, a low score means better outcome Externalizing problems score: range 0-70, a low score means better outcome
  Outcome analyses: Total syndrome scales at age 6 years.
BMI age 0-6 years | 6 years
  From parental reports every 6 months.
  Outcome analyses: development of BMI age 0-6 years and current BMI at age 6.
Waist circumference age 0-6 years | 6 years
  From parental reports every 6 months.
  Outcome analyses: development of waist circumference age 0-6 years and current waist circumference at age 6.
ADHD symptoms at age 3 years | 3 years
  From the ADHD rating scale-IV preschool, a dimensional questionnaire for ADHD symptoms in preschool children.
  For inattentive score: range: 0-27, a low score means better outcome. For impulsivity-hyperactivity: range: 0-27, a low score means better outcome.
  Outcome analyses: ADHD symptom scores at age 3 years.
Social behavior assessment at age 3 years | 3 years
  From the Social Responsiveness Scale, Second Edition; a questionnaire for screening for autistic traits:
  Total score range: 0-195, a low score indicates better outcome.
  Outcome analyses: Total problem scores at age 3 years.
Social behavior assessment at age 6 years | 6 years
  From the Social Responsiveness Scale, Second Edition; a questionnaire for screening for autistic traits.
  Total score range: 0-195, low score indicates a better outcome.
  Outcome analyses: Total problem scores at age 6 years.
Psychopathology screening at age 3 years | 3 years
  From the Child Behavior Check List 1,5-5 years; a questionnaire for general screening of preschool psychopathology.
  Total problem score: range 0-198, a low score means better outcome
  Outcome analyses: Total syndrome scales at age 3 years.
Adaptive behavior at 3 years | 3 years
  Adaptive Behavior Assessment System, Third Edition (ABAS-3)is used to assess everyday, adaptive functioning.
  Total score range: 0-645, a low score indicate poorer outcome.
Adaptive behavior at 6 years | 6 years
  Adaptive Behavior Assessment System, Third Edition (ABAS-3)is used to assess everyday, adaptive functioning.
  Total score range: 0-633, a low score indicate poorer outcome.
Cognitive assessment age 0-3 years | 3 years
  From Behavior Rating Inventory of Executive Function in preschool children; a measurement of executive functions.
  Total problem score: range 63-189, a low score means better outcome.
  Outcome analyses: Index values at age 3 years.
Cognitive assessment age 0-6 years | 6 years
  From Behavior Rating Inventory of Executive Function in preschool children; a measurement of executive functions.
  Total problem score: range 60-180, a low score means better outcome.
  Outcome analyses: Index values at age 6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, PhD, Principal Investigator — Copenhagen Studies on Asthma in Childhood; Bo Chawes, PhD, Principal Investigator — Copenhagen Studies on Asthma in Childhood
Locations (1):
- Copenhagen University Hospital of Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brustad N, Vahman N, Ralfkiaer U, Mikkelsen M, Brandt S, Kyvsgaard JN, Vinding R, Stokholm J, Chawes B, Bonnelykke K. Fish oil and vitamin D in pregnancy for the prevention of early childhood asthma: study protocol for two double-blinded, randomised controlled trials. BMJ Open. 2024 Dec 31;14(12):e092902. doi: 10.1136/bmjopen-2024-092902. PMID 39740942